CLINICAL TRIAL: NCT05702190
Title: Opium Tincture Against Chronic Diarrhea - Healthy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asbjørn Mohr Drewes (Other)
Responsible Party: Sponsor-Investigator, Asbjørn Mohr Drewes, Professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Dropizol_healthy; 2020-004875-41 (EudraCT Number)
Record Dates: First submitted 2023-01-06; First posted 2023-01-27 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Chronic Diarrhea
Keywords: Diarrhea; Constipation; Gastrointestinal transit
MeSH Terms: conditions — Diarrhea; Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opium tincture (Active Comparator): Administration of opium tincture (Dropizol)
  Interventions: Drug: Opium tincture
- Placebo (Placebo Comparator): Administration of placebo (identical to opium tincture in taste and appearance)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Opium tincture — Self-administration of opium tincture (10 mg/ml) as 2x5 drops on day 1, 3x10 drops on days 2-8, and 1x10 drops on day 9 in each study period.
  Other Names: Dropizol
  Arms: Opium tincture
Drug: Placebo — Self-administration of placebo as 2x5 drops on day 1, 3x10 drops on days 2-8, and 1x10 drops on day 9 in each study period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the mechanistic anti-propulsive effects of opium tincture on the gastrointestinal tract of a cohort of healthy participants.

DETAILED DESCRIPTION:
Opium tincture is used a symptomatic drug against chronic diarrhea even though no clinical studies have investigated the effect on gastrointestinal function. With this randomized, double-blind, placebo-controlled cross-over trial in 20 healthy participants, the investigators wish to provide evidence-based insights into the effects of opium tincture on gastrointestinal function. Additionally, effects on the central nervous system will be investigated a tertiary aim.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any study specific procedures
* Able to read and understand Danish
* Male or female with an age of 20 years or more
* The researcher believes that the participant understands what the study entails, are capable of following instructions, can attend when needed, and are expected to complete the study.
* The investigator will ensure that fertile female participants have a negative pregnancy test before each treatment visit and use contraception during the entity of the study.
* Opioid naïve (in this study "opioid naïve" is defined as a person who does not have a history of opioid use/addiction. If the opioids were used more than five years before the start of experiment as an analgesic to treat pain post-surgery etc., this person will be considered opioid naïve. If the person has never used opioids to treat pain but has participated in pain studies where opioids were given more than a year before this experiment, this person will be considered opioid naïve)
* Healthy (assessed by a study-affiliated medical doctor)

Exclusion Criteria:

* Known allergy towards pharmaceutical compounds similar to Dropizol.
* Participation in other studies within 14 days of first visit (1 year if opioids involved).
* Expected need of medical/surgical treatment during the study
* History of psychiatric illness (e.g. mental retardation, schizophrenia, affective disorders (depression), personality disorders or treatment with psychoactive medications)
* History of substance abuse (e.g. alcohol, nicotine, tetrahydrocannabinol (THC), benzodiazepine, central stimulants and/or opioids)
* Family history of substance abuse
* Known increased intracranial pressure
* Known major stenosis of the intestines
* Planned MRI within the next 3 months
* Metal implants or pacemaker
* Known severe decreased renal function (defined as estimated glomerular filtration rate (eGFR) below 45)
* Known severe decreased hepatic function (defined as Child-Pugh class B or higher)
* Treatment with Monoamine oxidase (MAO) inhibitors during the entity of the study
* Known severe chronic obstructive pulmonary disease (COPD) or acute severe asthma (defined as forced expiratory volume in 1 second (FEV1) below 50 % or acute ongoing exacerbation)
* Known cor pulmonale
* Female participants that are lactating
* Medicine known to affect gastrointestinal motility must not be initiated during the entity of the study
* Use of any analgesic medication within 48 hours before start as well as for the duration of the study (urine drug test will be performed prior to treatment start).
* Intake of alcohol within 48 hours before start of study period as well as for the duration of the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal transit | Measurement started on day 2 of each study period until expulsion of the capsule (typically 24-48 hours after)
  Difference in hours from ingestion of a 3D Transit Capsule to expulsion of the capsule during active and placebo treatment

SECONDARY OUTCOMES:
Colonic motility patterns | Measurement started on day 2 of each study period until expulsion of the capsule (typically 24-48 hours after)
  Number of motility patterns in the colon measured by the 3D Transit Capsule
Bowel movement frequency | From day 1 to day 9
  Number of spontaneous bowel movements per day
Stool consistency | From day 1 to day 9
  Rated on the Bristol Stool Form Scale (ranging from type 1 (constipation) - type 7 (diarrhea))
Pupil diameter | Day 1, 6, and 9
  Measured in mm
General cognition | Day 1, 6, and 9
  Evaluated using the Mini-Mental State Examination
Reaction time | Day 1, 6, and 9
  Measured in milliseconds (ms) from a sound was provided and until the participant pressed a button
Short-term memory | Day 1, 6, and 9
  Measured as number of digits correctly remembered after visual presentation
Gastrointestinal symptoms | Day 1-9
  Measured on the Gastrointestinal Symptom Rating Score (GSRS) questionnaire (ranging from 0 (no discomfort) to 6 (very severe discomfort)
Constipation symptoms | Day 1-9
  Measured on the Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire (ranging from 0 (symptom absent) to 4 (very severe).
Electroencephalography spectral analysis | Day 1 and 9
  40 electrodes will be used to record EEG during a period of 5 minutes rest. The results will be used to model connectivity between brain centres as well as the dominating centres of brain. EEG power will be assessed in the Delta, Theta, Alpha, Beta, and Gamma bands between 1 and 70 Hertz. Finally inverse modelling will be conducted to explore the dominating centres of brain activity.
Pain tolerance threshold | Day 1 and 9
  Pressure will be applied to the tibial bone and the quadriceps muscle by a handheld pressure algometer. The pain tolerance threshold (measured in kPa) is reached when the participant reports the pain to be intolerable
Conditioned pain modulation | Day 1 and 9
  The left hand of the participant is immersed in 2.0 degree (celsius) cold water for up to 2 minutes or until the pain becomes intolerable. The participant is asked to rate the pain on a 10-point Visual Analogue Scale (0 being no pain and 10 being worst imaginable pain) every 10 seconds during the test.
Gastric half emptying time | Day 1 and 9
  Analysis of gastric half emptying time after ingestion of a standardized meal measured by MRI
Gastric contraction assessment | Day 1 and 9
  Analysis of gastric contraction including amplitude and frequency of contractions after ingestion of a standardized meal measured by MRI
Small bowel motility assessment | Day 1 and 9
  Analysis of small bowel motility after ingestion of a standardized meal measured using dynamic MRI images. A semi-automated analysis software enables registration of small bowel motility with the calculation of regional motility maps and quantification of motility indices.
Small bowel water content | Day 1 and 9
  Analysis of small bowel water content measured using heavily T2-weighted MRI images
Colon volume | Day 1 and 9
  Volumetric quantification of the colon measured using T2-weighted MRI images
Estimated gastrointestinal transit time | Day 1 and 9
  Using DIXON images, location of three capsules filled with contrast fluid ingested 24 hours before MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Mohr Drewes, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data can by provided upon request
Access Criteria: Researchers who provide a methodological sound proposal